CLINICAL TRIAL: NCT06702631
Title: Functional MRI of Nitrous Oxide Inhalation in Volunteer Subjects
Brief Title: Nitrous Oxide Neuroimaging
Acronym: NONI
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Keith M Vogt (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Keith M Vogt, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY24100059; R35GM146822 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Pain; Amnesia
MeSH Terms: conditions — Pain; Amnesia | interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Nitrous Oxide + Pain (Experimental): Single-arm study. All subjects receive nitrous oxide and painful electric nerve stimulation, as described in the interventions.
  Interventions: Drug: Nitrous oxide; Device: Peripheral Nerve Stimulation

INTERVENTIONS:
Drug: Nitrous oxide — After a no-drug control period, subjects will inhale nitrous oxide, administered via a breathing circuit and face mask, until a steady-state target end-tidal expired concentration is reached. During the drug condition, subjects will receive low-dose nitrous oxide (% corresponding to Minimum Alveolar Concentration).
Device: Peripheral Nerve Stimulation — Experimental acute pain stimulus will be delivered using a nerve stimulator. These painful shocks will be paired with a fixed number of the experimental cues, in a pattern that appears random to participants.

SUMMARY:
The purpose of this study is to determine the effects of acute pain on long-term memory and conditioned physiologic responses in the presence and absence of low dose nitrous oxide. Functional magnetic resonance imaging will be used to identify the neural correlates of these phenomena. The study will occur over 2 visits and involves no long-term follow up.

DETAILED DESCRIPTION:
This is a non-randomized, clinical trial study of healthy volunteer subjects, which will employ neuroimaging and behavioral measures to characterize the effects of inhalational nitrous oxide on pain processing and cognitive function. Sedative doses of nitrous oxide will be targeted, and steady-state end-tidal (expired) concentrations achieved, while subjects perform a pain and memory cognitive task. At both no-drug baseline and the targeted doses, task and resting-state functional magnetic resonance imaging (MRI) scans will be acquired, and this data will be analyzed subsequently for task-related brain activity (from pain processing and memory formation) and functional connectivity. This work will use a systems neuroscience approach to fill an important knowledge gap about the central effects of inhalational nitrous oxide in the context of painful stimulation.

The investigators propose to complete the following 3 Aims, at a targeted sedative dose of nitrous oxide, compared to no-drug baseline, using functional MRI:

Aim 1: Determine how the brain response to acute pain stimulation is modulated by nitrous oxide. It is anticipated that nitrous oxide will correlate to decreased activation in both somatosensory (thalamus, insula, primary somatosensory/motor) and affective (anterior cingulate) components of the pain processing brain areas.

Aim 2: Determine how memory encoding is modulated by nitrous oxide, in the context of periodic painful stimulation. It is anticipated that nitrous oxide will correlate to decreased activation in both the explicit memory (hippocampus, parahippocampus) and associative learning (amygdala, anterior cingulate) brain systems.

Aim 3: Determine the neural effects of inhalational nitrous oxide on brain connectivity both at rest and during the combined pain and memory task performance. It is anticipated that nitrous oxide will cause widespread dose-dependent decreases in long-range functional connectivity between brain areas known to be involved in pain processing and to the default mode network, and that this connectivity will differ between the resting (task-free) and periodic pain states.

ELIGIBILITY:
Inclusion Criteria:

* have none of the specific exclusion criteria
* have a valid email address and valid phone number throughout the study
* free from any non-MRI compatible implants

Exclusion Criteria:

* are pregnant or attempting to conceive
* body mass index (BMI) > 35
* significant memory impairment or hearing loss
* sleep apnea
* chronic pain or frequently taking pain medication (including tramadol)
* any severe or poorly-controlled medical problem (hypertension, diabetes)
* neurologic or psychiatric disease, including anxiety, and depression
* severe cardiac disease
* history of methylenetetrahydrofolate reductase (MTHFR) deficiency or variant mutation, as assessed by personal report
* recent ear or eye surgery
* being claustrophobic
* have metal implants or non-removable metal piercings
* having a history of adverse reaction to anesthetics
* daily alcohol or heavy alcohol use; history of alcohol abuse
* current daily smoker
* regular or recent marijuana use (including prescribed/medical marijuana)
* illicit drug use, i.e., street drugs
* regularly taking: antiepileptics, antidepressants, anti-psychotics, antihistamines, anti-anxiety medication, stimulants, or sleep-aids

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Brain activation to painful stimulation difference: Drug-free condition minus nitrous oxide condition | Visit 1: Immediate; average activity, calculated from each task scan
  Event-related blood-oxygen level dependent Magnetic Resonance Imaging (MRI) responses will be determined. Z-scores will be calculated by linear regression of the task timing against the MRI signal time-course (MRI data is in arbitrary units with no maximum or minimum) at each voxel (single data point in brain). Primary outcome will be for the right insula. Z-score of 0 indicates no task-related changes. Z-scores further from zero indicate stronger correlation between functional MRI signal change and the task timing, with positive values indicating increases in functional MRI signal and negative Z-scores indicating decreases. Practically, higher positive Z-scores would indicate increased brain activity and larger negative Z-scores would indicate decreased brain activity.
Resting-state functional connectivity difference: Drug-free minus nitrous oxide condition | Visit 1: Immediate; brain activity captured in data acquired across entire 6-8 minute scan.
  Functional connectivity (FC) will be calculated as the correlation between the time-series of MRI signal (MRI data is in arbitrary units with no maximum or minimum) on a pair-wise basis between every atlas-defined region in the brain. Strength of temporal correlation is reflective of brain regions that are working together, and changes in FC reflect differences in brain state, in this case between the drug-free and nitrous oxide conditions. The reported value will be for FC change between insula and anterior cingulate. T-score of 0 would indicate no condition-related changes in connectivity between the two brain regions. T-scores further from zero indicate stronger connectivity change: positive T-score reflects drug-free > nitrous oxide; negative T-scores indicate nitrous oxide > drug-free.

SECONDARY OUTCOMES:
Explicit memory performance | Visit 2: 24 hours post-learning experiment
  Recognition memory testing, using the Remember-Know procedure, in which subjects indicate whether they recognize previously experienced experimental items among novel items (not previously in the experiment). This allows calculation of interdependent measures of recollection & familiarity using the signal detection statistic, d'. d' is calculated as the cumulative Gaussian distribution of false positive responses subtracted from the cumulative Gaussian distribution of correctly identified previously-experienced items. d' is on a (theoretically infinite) scale of standard deviation units, with negative values representing performance worse than chance guessing and positive values representing stand deviations of performance above chance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data to share:
  * age, height, weight, sex
  * survey instruments to quantify pain predispositions (catastrophizing, vigilance & anxiety), depression, anxiety, stress, and sleep
  * pain intensity & unpleasantness, and observer assessment of sedation at the targeted drug dose
  * Behavioral performance data for long-term memory
  * structural and functional magnetic resonance images
Supporting Information: Study Protocol
Time Frame: After analysis is complete and results have been published, all the above data will be shared in de-identified format, linked together by an assigned subject number.
Access Criteria: Data will be shared via a publicly-accessible online platform that allows user download at no cost.